CLINICAL TRIAL: NCT04598984
Title: The Role of Serum Adipokines in Predicting Response to Neoadjuvant Therapy in Patients With Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cihad Tatar, Associate Profesor, Istanbul Training and Research Hospital
Other Study IDs: 2506
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer Stage III
Keywords: rectal cancer; neoadjuvant; serum adipokines; leptin; adiponectin
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low levels of serum adipokines
  Interventions: Diagnostic Test: serum adipokines
- High levels of serum adipokines
  Interventions: Diagnostic Test: serum adipokines

INTERVENTIONS:
Diagnostic Test: serum adipokines — Level of serum adipokines will be measured with flow cytometry

SUMMARY:
It has been shown that adipokines (resistin, leptin, adiponectin) secreted from adipose tissue and proinflammatory cytokines such as IL-6, TNF-a are associated with the risk of developing colorectal cancer. However, the role of these factors in predicting clinical response to neoadjuvant therapy in rectal cancers is unknown. In this study, the role of serum adipokine levels before neoadjuvant therapy in predicting clinical response in patients with rectal cancer is investigated. For this purpose, blood will be drawn from patients with rectal cancer who will receive neoadjuvant therapy, serum adipokines will be studied and clinical response to neoadjuvant therapy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients with locally advanced rectal cancer

Exclusion Criteria:

* below 18 years old
* patients who did not received neoadjuvant therapyAll

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with locally advanced rectal cancer
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The Role of Serum Adipokines in Predicting Response to Neoadjuvant Therapy in Patients with Rectal Cancer | 1 year
  The Adiponectin, Adipsin, Leptin, Resistin levels will be measured with flow cytometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided